CLINICAL TRIAL: NCT00739089
Title: A Pilot Study to Compare the Interaction Between Central Venous Mixed Venous Oxygen Saturation Catheters and Central Venous Hemodialysis Catheters
Brief Title: Presep and Vascath Interaction Study
Status: Withdrawn | Type: Observational
Why Stopped: Study stopped due to a lack of enrollment.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00004073
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-01

CONDITIONS: Hemodynamics; Renal Dialysis; Sepsis; Shock
Keywords: hemodynamics; oxygen; renal dialysis; shock; sepsis; hypotension; lactic acidosis
MeSH Terms: conditions — Sepsis; Shock; Hypotension; Acidosis, Lactic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, observational study to compare presep(tm) catheter central vein mixed venous oxygen saturation before and after dialysis is initiated via the vascath(tm) central venous dialysis catheter to evaluate device interaction.

DETAILED DESCRIPTION:
The central venous oxygen saturation catheter measurement may be influenced by close approximation to the tip of the central venous hemodialysis catheter when hemodialysis is ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the MICU
* PreSep venous oxygen saturation central venous catheter already in place
* VasCath central venous dialysis catheter already in place
* Planned hemodialysis

Exclusion Criteria:

* Patient unable to undergo hemodialysis
* Contraindication for PreSep or VasCath catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: medical intensive care unit (MICU) patients in an academic tertiary care referral medical center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
change in SvO2 | before and afer initiation of dialysis via a vascath

CONTACTS AND LOCATIONS:
Overall Officials: Arjun B Chatterjee, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data would have been shared with any other investigator with a local IRB approved protocol to evaluate de-identified patient data

REFERENCES:
- [Background] Vaziri ND, Wilson A, Mukai D, Darwish R, Rutz A, Hyatt J, Moreno C. Dialysis hypoxemia. Role of dialyzer membrane and dialysate delivery system. Am J Med. 1984 Nov;77(5):828-33. doi: 10.1016/0002-9343(84)90519-9. PMID 6496536
- [Background] Jakob SM, Ruokonen E, Vuolteenaho O, Lampainen E, Takala J. Splanchnic perfusion during hemodialysis: evidence for marginal tissue perfusion. Crit Care Med. 2001 Jul;29(7):1393-8. doi: 10.1097/00003246-200107000-00015. PMID 11445693
- [Background] Krafft P, Steltzer H, Hiesmayr M, Klimscha W, Hammerle AF. Mixed venous oxygen saturation in critically ill septic shock patients. The role of defined events. Chest. 1993 Mar;103(3):900-6. doi: 10.1378/chest.103.3.900. PMID 8449089
- [Background] De Backer WA, Verpooten GA, Borgonjon DJ, Vermeire PA, Lins RR, De Broe ME. Hypoxemia during hemodialysis: effects of different membranes and dialysate compositions. Kidney Int. 1983 May;23(5):738-43. doi: 10.1038/ki.1983.87. No abstract available. PMID 6876569
- [Background] Quebbeman EJ, Maierhofer WJ, Piering WF. Mechanisms producing hypoxemia during hemodialysis. Crit Care Med. 1984 Apr;12(4):359-63. doi: 10.1097/00003246-198404000-00004. PMID 6705543
- [Background] Murray P, Hall J. Renal replacement therapy for acute renal failure. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):777-81. doi: 10.1164/ajrccm.162.3.ncc400. No abstract available. PMID 10988080